CLINICAL TRIAL: NCT02159469
Title: A Multiple-dose, 52-week Study to Evaluate the Efficacy and Safety of Testosterone Enanthate Administered Subcutaneously Once Each Week to Adult Males With Hypogonadism
Brief Title: Subcutaneous Testosterone Replacement Efficacy and Safety in Adult Men Diagnosed With Hypogonadism
Acronym: STEADY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QST-13-003
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone enanthate
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone enanthate auto-injector (Experimental): Testosterone enanthate 50 mg / 75 mg / 100 mg administered subcutaneously once each week with possible titration to a higher or lower dose at scheduled intervals during study.
  Interventions: Combination Product: Testosterone enanthate auto-injector

INTERVENTIONS:
Combination Product: Testosterone enanthate auto-injector — Dose Adjustment to 50 mg or 75 mg or 100 mg based upon Testosterone levels
  Other Names: Testosterone; Testosterone enanthate; QuickShot® Testosterone (QST)

SUMMARY:
Evaluation of efficacy and safety of testosterone enanthate administered subcutaneously using an auto-injector

DETAILED DESCRIPTION:
This study will evaluate, if testosterone enanthate administered subcutaneously once each week by an auto-injector to men with low testosterone, can raise their levels into the normal range.

The study will investigate the ability to adjust testosterone enanthate dose levels using single point blood concentrations.

Safety and tolerability of testosterone administration will be evaluated along with the patient's ability to use the auto-injector and follow the instructions for auto-injector use.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged ≥ 18 year of age with a documented diagnosis of hypogonadism
* Total testosterone levels < 300 ng/dL at two qualification visits
* Patients in good general health

Exclusion Criteria:

* Allergy to sesame or testosterone products
* BMI ≥ 40 kg/m2
* Hematocrit ≥ 52%
* History or current evidence of breast or prostate cancer
* Elevated PSA (Prostate-Specific Antigen) for age.
* Abnormal DRE (digital rectal examination)
* Obstructive uropathy of prostatic origin
* Poorly controlled diabetes
* Congestive heart failure
* Within 6 months of screening, MI (myocardial ischemia), unstable angina leading to hospitalization, percutaneous coronary intervention, coronary artery bypass graft, uncontrolled cardiac arrhythmia, stroke transient ischemia attack, ceratoid revascularization, endovascular procedure, or surgical intervention for peripheral vascular disease.
* History or current treatment of thromboembolic disease.
* Use of ACTH (adrenocorticotropic hormone) or oral/depot corticosteroids within 6 weeks of screening.
* History of severe, untreated sleep apnea
* Subjects with any clinically significant medical condition which, in the opinion of the investigator, would make the subject an unsuitable candidate for enrollment in the study
* Positive serology for HIV, hepatitis B or hepatitis C
* Current evidence of drug or alcohol abuse.
* Skin conditions in injection site that could confound injection site assessments.
* Administration of other investigational compounds within one month of screening or 5 half-lives of the investigational compound, whichever is longer).
* Use of estrogen, GnRH (gonadotropin-releasing hormone) or growth hormone within 12 months of screening.
* Use of other androgens (DHEA(Dehydroepiandrosterone), anabolic steroids, other sex hormones) or other substances/supplements know to affect the PK (pharmacokinetics) of testosterone enanthate
* Considered or scheduled surgical or dental procedures associated with blood loss ≥500 mL during study.
* Donation of plasma or blood within 56 days of screening or history of donation of > 50 mL of blood or plasma within 3 months of screening.
* Donation of plasma or blood during study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed Kaminetsky, MD, Principal Investigator — Manhattan Medical Research Practice
Locations (28):
- United States (28):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tucson, Arizona
  - Burbank, California
  - Torrance, California
  - Upland, California
  - Jacksonville, Florida
  - Oviedo, Florida
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Brookline, Massachusetts
  - Methuen, Massachusetts
  - Kansas City, Missouri
  - Lawrenceville, New Jersey
  - Albany, New York
  - New York, New York
  - Rochester, New York
  - Franklin, Ohio
  - Medford, Oregon
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas
  - Sugar Land, Texas
  - West Valley City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 150 patients were enrolled in this study. 128 patients completed through at least Week 26, 98 patients completed through Week 52, and 97 patients completed the full study (through the Follow-up Visit).
Pre-assignment Details: The study was designed to ensure a minimum of 100 patients completed a collection of 26 weeks of safety data, and a minimum of 50 patients completed a collection of 52 weeks of safety data. Minimum enrollment goals were exceeded.
Groups:
- QST 50 mg / 75 mg / 100 mg: Testosterone enanthate 50 mg / 75 mg / 100 mg dose administered subcutaneously once each week with possible titration to a higher or lower dose at scheduled intervals during study.
Period: Overall Study
Arm/Group | QST 50 mg / 75 mg / 100 mg
Started | 150
Completed 12 Week | 137
Completed | 97
Not Completed | 53
Not completed — Missing Completion status | 1
Not completed — Adverse Event | 5
Not completed — Non-compliance | 2
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Sponsor's request | 2
Not completed — Met Stopping Criteria | 3
Not completed — Other | 1
Not completed — Multiple | 29

BASELINE CHARACTERISTICS:
Population: Masked dose assignment based upon Testosterone levels; Individual patients may receive all three dose levels.
Groups:
- Testosterone Enanthate Auto-injector: Testosterone enanthate administered subcutaneously once each week with possible titration to a higher or lower dose at scheduled intervals during study.
  Testosterone enanthate auto-injector Dose Adjustment: 50 mg / 75 mg / 100 mg
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 142
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 133
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Total Testosterone Cavg(0-168h) Serum Concentrations Within the Normal Range (300-1100 ng/dL)
Description: The primary objective of this study was to demonstrate the efficacy of QST (QuickShot Testosterone) administered subcutaneously once each week to adult males with hypogonadism.
Time Frame: 12 weeks
Population: The Population consisted of all patients who received at least 1 dose of the investigational product. Percentage was calculated using the number of patients in the column heading as the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 150
Participants | 139

2. Secondary Outcome: Safety and Tolerability
Description: * Incidence of adverse events throughout the study
  * Incidence and severity of injection site reactions throughout the study
Time Frame: 52 weeks
Population: TEAE (Treatment-emergent adverse event)s were defined as any event that started on or after the first dosing of IP (Investigational Product), or existed prior to the first dose and worsened in severity or relatedness to IP after dosing. The Population consisted of all patients who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Testosterone Enanthate Auto-injector: Testosterone enanthate administered subcutaneously once each week with possible titration to a higher or lower dose at scheduled intervals during study.
  Testosterone enanthate auto-injector Dose Adjustment 50 mg / 75 mg / 100 mg
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 150
Participants
  Patients with any TEAE | 125
  Patients with any TEAE related to IP | 66
  Patients with any SAE | 3
  Patients with TEAE leading to discontinuation | 30
  Patients discontinued due to IP related TEAE | 1
  Patients with any adverse event leading to death | 1

ADVERSE EVENTS:
Time Frame: Incidence of Adverse Events Throughout the Study, During the 12-Week Titration Phase, and During the Extended Treatment Phase up to 52 weeks
Description: Treatment-emergent adverse events were defined as any event that started in the study on or after the first dosing of IP, or existed prior to the first dose and worsened in severity or relatedness to IP after dosing. Percentage was calculated using the number of patients in the column heading as the denominator.
  In total, 125 (83.3%) patients had TEAEs during the study.
Arm/Group | Testosterone Enanthate Auto-injector
All-Cause Mortality (participants affected / at risk) | 1/150
Serious Adverse Events (participants affected / at risk) | 3/150
Other Adverse Events (participants affected / at risk) | 125/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate Auto-injector (N=150)
Depression (Psychiatric disorders) | 1 (1) — Worsening depressive disorder
Suicide (Psychiatric disorders) | 1 (1) — SUICIDE, METHOD UNKNOWN
Vertigo (Ear and labyrinth disorders) | 1 (1) — Vertigo
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate Auto-injector (N=150)
Hematocrit increased (Investigations) | 21 (21)
Prostatic specific antigen increased (Investigations) | 18 (18)
Blood creatine phosphokinase increased (Investigations) | 5 (5)
Blood testosterone increased (Investigations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 12 (12)
Sinusitis (Infections and infestations) | 11 (11)
Nasopharyngitis (Infections and infestations) | 6 (6)
Bronchitis (Infections and infestations) | 5 (5)
Influenza (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Injection site bruising (General disorders) | 10 (10)
Injection site hemorrhage (Gastrointestinal disorders) | 5 (5)
Injection site erythema (General disorders) | 4 (4)
Edema peripheral (General disorders) | 4 (4)
Fatigue (General disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 19 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (8)
Prostatitis (Reproductive system and breast disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 3 (3)
Polycythemia (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other